CLINICAL TRIAL: NCT03172819
Title: An Open Label Phase I Study to Evaluate the Safety and Efficacy of OBP-301 With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: Special Combination of OBP-301 and Pembrolizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toshihiko Doi (Other)
Collaborators: Oncolys BioPharma Inc (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Toshihiko Doi, Chief / Division of experimental therapeutics, National Cancer Center Hospital East
Organization: National Cancer Center Hospital East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC1505
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OBP-301+Pembrolizumab (Experimental): OBP-301+Pembrolizumab
  Interventions: Biological: OBP-301; Drug: Pembrolizumab

INTERVENTIONS:
Biological: OBP-301 — Intratumoral injection directly into the dose target region of a tumor at Day 1, Day 15, and Day 29.
  Additional administration of OBP-301 After the recommended dose of OBP-301 has been established, additional administration of OBP-301 is allowed. After completion of administration of OBP-301 on Day 1 - Day 29(+/- 4 days), if the target region has not disappeared, additional administration of OBP-301 is allowed after Day 43 or later.
  The patients in Phase 1a, Pembrolizumab administration has continued, are included.
  The recommended dose determined in the Phase 1a part will be administered 3 times biweekly (+/- 4 days); max 4 cycles.
Drug: Pembrolizumab — 200 mg Pembrolizumab is infused intravenously at Day 8. Thereafter infusion will continue every 3 weeks until discontinuation.

SUMMARY:
This is multicenter, open-label Phase I study to exploratively evaluate the efficacy and safety of OBP-301 in combination with Pembrolizumab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Phase 1a part:

To evaluate safety and tolerability in combination of OBP-301 and Pembrolizumab in patient with advanced or metastatic solid tumor and to determine recommended dose in phase 1b part.

Phase 1b part:

To evaluate safety and potential efficacy in combination of OBP-301 and Pembrolizumab in patients in expanded arm.

ELIGIBILITY:
Inclusion criteria

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >=18 years of age on the day of signing the informed consent.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Have histologically or cytologically confirmed advanced or metastatic solid tumor with possibility of intratumoral injection, for which no effective standard therapy exists or standard therapy has failed.
5. Have one or more evaluable lesions based on RECIST 1.1

   *Evaluable lesions: measurable lesion and/or non-measurable lesion
6. Be willing to provide tissue; newly obtained endoscopic biopsy specimens or formalin-fixed, paraffin-embedded (FFPE) block specimens.
7. Female subjects of childbearing potential have a negative urine or serum pregnancy test within 7 days prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. It is allowed that the test at the same day at 7 days prior to enrollment. And male / female subjects of childbearing potential must be agree to use an adequate method of contraception starting with signing the informed consent through 120 days after the last dose of study medication.
8. Demonstrated adequate organ function as defined in following criteria. All screening labs should be performed within 7 days of enrollment. It is allowed that the labs at the same day at 7days prior to enrollment.

Note: Subject must not have taken transfusion, hematopoietic agent; granulocyte-colony stimulating factor (G-CSF) etc., and/or oxygen inhalation within 7 days before the screening labs.

1. Absolute neutrophil count (ANC)>=1,500 /mm3
2. Platelets>=100,000 /mm3
3. Hemoglobin>=9.0 g/dL
4. Serum total bilirubin<=2.0 mg/dL
5. aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT)<=100 IU/L for subjects with liver metastases<=200 IU/L
6. Serum creatinine<= 1.5 mg/dL; or if serum creatinine > 1.5 mg/dL, creatinine/clearance >=60 mL/min (Cockcroft-Gault formula)

Exclusion criteria

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of study Day 1.
2. Has an active autoimmune disease that has required systemic treatment in past 2 years.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study Day 1.
4. Has known active central nervous system metastases and/or carcinomatous meningitis.
5. Has had prior anti-cancer monoclonal antibody chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or immunotherapy targeted to Programmed cell death 1 (PD-1), PD-L1, PD-L2 within 4 weeks prior to Da y 1 or OBP-301 study, who has not recovered from adverse events due to a previously administered agent.
6. Has a known additional malignancy that is progressing or requires active treatment.
7. Has received a live vaccine within 30 days of planned start of study therapy.
8. Has a known history of Human Immunodeficiency Virus.
9. Has known active Hepatitis B or Hepatitis C.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
14. Previous severe hypersensitivity to another monoclonal antibody
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 4weeks
  Dose limiting toxicity

SECONDARY OUTCOMES:
Response rate (RR) | 3 years
  Response rate by RECIST ver. 1.1
Progression free survival (PFS) | 3 years
  Progression free survival
Rate of adverse event | 3 years
  Rate of adverse event

OTHER OUTCOMES:
Biomarkers:Efficacy evaluations according to immune status | 3 years
  Immune status will be analyzed using biopsy and blood samples by flow cytometry, RNA seq, whole exome sequencing, and immunohistochemistry, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiko Doi, Dr, Study Chair — National Cancer Center Hospital East
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No